CLINICAL TRIAL: NCT01711632
Title: A Phase II Study of the BRAF Inhibitor, Vemurafenib, in Patients With Relapsed or Refractory Hairy Cell Leukemia
Brief Title: BRAF Inhibitor, Vemurafenib, in Patients With Relapsed or Refractory Hairy Cell Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Northwestern University (Other); Ohio State University (Other); Dana-Farber Cancer Institute (Other); Scripps Clinic (Other); Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-200
Record Dates: First submitted 2012-10-17; First posted 2012-10-22 (Estimated); Results first posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2024-08

CONDITIONS: Hairy Cell Leukemia
Keywords: VEMURAFENIB; BRAF Inhibitor; 12-200; Zelboraf™
MeSH Terms: conditions — Leukemia, Hairy Cell | interventions — Vemurafenib

ARMS (1):
- Vemurafenib (Experimental): Eligible patients will receive vemurafenib at a dose of 960mg orally twice daily (b.i.d.) continuously in cycles of 4 weeks (28 days).
  Interventions: Drug: Vemurafenib

INTERVENTIONS:
Drug: Vemurafenib — Patients will receive vemurafenib at a dose of 960mg orally b.i.d. continuously in cycles of 4 weeks (28 days) as outpatient. A bone marrow aspirate and/or biopsy will be performed after the first cycle for research purposes only. After the completion of the third cycle, a repeat bone marrow aspirate and/or biopsy will be performed for assessment of response and evaluation of MRD. Following the third cycle assessments, patients who achieve complete response (CR) with detectable MRD or partial response (PR) may continue with vemurafenib for up to 3 additional cycles at the treating physician's discretion (Cycles 4-6). Patients who achieve CR without MRD will be observed as part of post-treatment followup, and may be re-treated with vemurafenib after relapse (as per below). Patients who achieve no response (NR) after the initial 3 cycles of vemurafenib will be removed from the study. They will be followed every 3 months as part of posttreatment followup for a total of 12 months.
  Other Names: Zelboraf™

SUMMARY:
The purpose of this study is to find out what effects, good and/or bad, treatment with vemurafenib (also known as Zelboraf™) has on the patient and on leukemia. Specifically, the researchers want to know how well vemurafenib eliminates leukemia from the blood.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Histologically confirmed classical HCL with one of the following:
* Intolerance to purine analogs or considered to be poor candidates for purine analog-based therapy
* Failure to achieve any response (CR or PR) to the initial purine analog-based therapy
* Relapse ≤ 2 years of purine analog-based therapy
* ≥ 2 relapses Histologic confirmation of diagnosis will be performed at MSKCC or a participating site.
* Patients who meet the standard treatment initiation criteria, as defined by ANC ≤1.0, Hgb ≤ 10.0 or PLT ≤100K
* ECOG performance status of 0-2
* Acceptable pre-study organ function during screening as defined as: Total bilirubin ≤ 1.5 times the upper limit of normal (ULN), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5x ULN, and serum creatinine ≤ 1.5x ULN
* Electrocardiogram (ECG) without evidence of clinically significant ventricular arrhythmias or ischemia as determined by the investigator and a rate-corrected QT interval (QTc, Bazett's formula) of < 480 msec.
* For women of childbearing potential, agreement to the use of two acceptable methods of contraception, including one barrier method, during the study and for 6 months after discontinuation of vemurafenib
* For men with female partners of childbearing potential, agreement to use a latex condom and to advise their female partner to use an additional method of contraception during the study and for 6 months after discontinuation of vemurafenib
* Negative serum pregnancy test within 7 days of commencement of treatment in premenopausal women.
* Agreement not to donate blood or blood products during the study and for at least 6 months after discontinuation of vemurafenib; for male partners, agreement not to donate sperm during the study and for at least 6 months after discontinuation of vemurafenib
* Ability to understand and willingness to sign a written informed consent document.
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

* Pregnant or breast-feeding
* Have had chemotherapy (including purine analogs, rituximab, and other investigational agents) within six weeks prior to entering the study
* Major surgery within 4 weeks prior to entering the study
* Invasive malignancy within the past 2 years prior to first study drug administration, except for adequately treated (with curative intent) basal or squamous cell carcinoma, melanoma, in situ carcinoma of the cervix, in situ ductal adenocarcinoma of the breast, in situ prostate cancer, or limited stage bladder cancer or other cancers from which the patient has been disease-free for at least 2 years
* Refractory nausea or vomiting, malabsorption, external biliary shunt, or history of any type of gastrointestinal surgery that would preclude adequate absorption of study drug
* Prior treatment with MEK or BRAF inhibitors
* Active HIV, hepatitis B and hepatitis C
* Patients with HCL variant (as defined by absence of expression of CD25 or absence of BRAF V600E mutation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2024-08-16 (Actual); Study Completion 2024-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jae H. Park, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Scripps Clinic, La Jolla, California
  - Northwestern University, Evanston, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Ohio State University, Columbus, Ohio

REFERENCES:
- [Derived] Handa S, Lee JO, Derkach A, Stone RM, Saven A, Altman JK, Grever MR, Rai KR, Shukla M, Vemuri S, Montoya S, Taylor J, Abdel-Wahab O, Tallman MS, Park JH. Long-term outcomes in patients with relapsed or refractory hairy cell leukemia treated with vemurafenib monotherapy. Blood. 2022 Dec 22;140(25):2663-2671. doi: 10.1182/blood.2022016183. PMID 35930750
- [Derived] Tiacci E, Park JH, De Carolis L, Chung SS, Broccoli A, Scott S, Zaja F, Devlin S, Pulsoni A, Chung YR, Cimminiello M, Kim E, Rossi D, Stone RM, Motta G, Saven A, Varettoni M, Altman JK, Anastasia A, Grever MR, Ambrosetti A, Rai KR, Fraticelli V, Lacouture ME, Carella AM, Levine RL, Leoni P, Rambaldi A, Falzetti F, Ascani S, Capponi M, Martelli MP, Park CY, Pileri SA, Rosen N, Foa R, Berger MF, Zinzani PL, Abdel-Wahab O, Falini B, Tallman MS. Targeting Mutant BRAF in Relapsed or Refractory Hairy-Cell Leukemia. N Engl J Med. 2015 Oct 29;373(18):1733-47. doi: 10.1056/NEJMoa1506583. Epub 2015 Sep 9. PMID 26352686
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vemurafenib
Started | 36
Completed | 14
Not Completed | 22
Not completed — Adverse Event | 4
Not completed — Death | 3
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 4
Not completed — Progressive disease | 2
Not completed — No follow up required in re-treatment | 3
Not completed — No follow up required in re-treatment | 3

BASELINE CHARACTERISTICS:
Arm/Group | Vemurafenib
Number analyzed (Participants) | 36
Age, Continuous [Median (Full Range); unit: years] | 60 [34 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 33
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Vemurafenib
Description: as assessed by overall response rates after three months of treatment in patients with relapsed or refractory HCL. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Vemurafenib
Number analyzed (Participants) | 36
Participants
  Complete Response | 10
  Partial Response | 14
  No CR or PR | 12

2. Secondary Outcome: Toxicity (Safety and Tolerability)
Description: Toxicity will be graded and recorded using the NCI Common Toxicology Criteria version 4.0.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Vemurafenib
Number analyzed (Participants) | 36
Participants
  Dose reduction to 720mg twice daily | 2
  Dose reduction to 480mg twice daily | 10
  Dose reduction to 240mg twice daily | 1
  Did not need a dose reduction | 23

3. Secondary Outcome: To Assess the Pharmacodynamics Change From Baseline
Description: Peripheral blood and/or bone marrow aspirate samples from pretreatment and post-treatment at specified time points will be assessed by Western Blot or by phospho-flow for the downstream targets of BRAF (MEK, pMEK, ERK, pERK) to assess the ontarget effect of the Vemurafenib. The droplet digital PCR assay was performed to quantify the concentration of molecules with mutated BRAF V600E DNA at baseline and again at 12 weeks of vermurafenib therapy.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Vemurafenib
Number analyzed (Participants) | 36
participants
  Pts with a decrease of the concentration of molecules with mutated BRAF V600E DNA at 12 wks | 24
  Pts without decrease of the concentration of molecules with mutated BRAF V600E DNA at 12 wks | 12

4. Secondary Outcome: Evaluate Biomarkers of Resistance
Description: Reactivation of MAPK pathways: Increased expression of the other RAF isoforms CRAF and ARAF), and MAPK (MAPK8 or COT) will be analyzed by Western Blot and/or real-time PCR39,40. Secondary BRAF mutations (all 18 BRAF exons) and RAS mutations40 will be analyzed by bidirectional Sanger sequencing and by Raindance multiplex PCR and Illumina next generation sequencing, respectively. Activation of RTKs (i.e. PDGFRβ and IGF-IR) will be assessed by Western Blot. Cell Biosciences NanoPro 1000 technology will be used to examine quantitative signaling on the entire MAPK, PI3K and JAK-STAT pathways41.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Vemurafenib
Number analyzed (Participants) | 36
Participants
  Participants with KRAS mutations | 1
  Participants without KRAS mutations | 35

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Vemurafenib
All-Cause Mortality (participants affected / at risk) | 7/36
Serious Adverse Events (participants affected / at risk) | 13/36
Other Adverse Events (participants affected / at risk) | 22/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vemurafenib (N=36)
Abdominal pain (Gastrointestinal disorders) | 1
Anaphylaxis (Immune system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Blood bilirubin increased (Investigations) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 5
Fever (General disorders) | 3
Gastrointestinal disorders, other (Gastrointestinal disorders) | 1
Hematoma (Vascular disorders) | 1
Lung infection (Infections and infestations) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Rectal hemorrhage (Gastrointestinal disorders) | 1
Skin & subcutaneous tissue disorders, other (Skin and subcutaneous tissue disorders) | 1
Syncope (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vemurafenib (N=36)
Hyperglycemia (Metabolism and nutrition disorders) | 21
Platelet count decreased (Blood and lymphatic system disorders) | 21
Anemia (Blood and lymphatic system disorders) | 20
Neutrophil count decreased (Investigations) | 19
White blood cell decreased (Investigations) | 19
Lymphocyte count decreased (Investigations) | 17
Blood bilirubin increased (Investigations) | 14
Alkaline phosphatase increased (Investigations) | 12
Alanine aminotransferase increased (Investigations) | 11
Hypoalbuminemia (Metabolism and nutrition disorders) | 10
Aspartate aminotransferase increased (Investigations) | 9
Creatinine increased (Investigations) | 8
Hypocalcemia (Metabolism and nutrition disorders) | 8
Hypophosphatemia (Metabolism and nutrition disorders) | 8
Hypernatremia (Metabolism and nutrition disorders) | 7
INR increased (Investigations) | 7
Hyponatremia (Metabolism and nutrition disorders) | 6
Hyperkalemia (Metabolism and nutrition disorders) | 5
Activated partial thromboplastin time prolonged (Investigations) | 4
Hypoglycemia (Metabolism and nutrition disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 3
Fibrinogen decreased (Investigations) | 1
Hemoglobin increased (Investigations) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-15): https://cdn.clinicaltrials.gov/large-docs/32/NCT01711632/Prot_SAP_000.pdf